CLINICAL TRIAL: NCT03133715
Title: Laparoscopic Versus Robot-assisted Ventral Hernia Repair: The Immediate, Intermediate, and Long Term Outcome Differences. A Single Institution Randomized Controlled Trial
Brief Title: Laparoscopic Versus Robot-assisted Ventral Hernia Repair: a Single Institution Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not IRB approved.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601533
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-06

CONDITIONS: Ventral Hernia
Keywords: robot-assisted
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either laparoscopic or robot-assisted repair of ventral hernia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic ventral hernia (Active Comparator): laparoscopic ventral hernia repair
  Interventions: Procedure: laparoscopic repair
- robot-assisted ventral hernia (Active Comparator): robot-assisted ventral hernia repair
  Interventions: Procedure: robot-assisted repair

INTERVENTIONS:
Procedure: laparoscopic repair — surgical repair of ventral hernia using laparoscopic repair
  Arms: laparoscopic ventral hernia
Procedure: robot-assisted repair — surgical repair of ventral hernia using robot-assisted repair
  Arms: robot-assisted ventral hernia

SUMMARY:
Randomized trial to compare outcomes of robot-assisted and laparoscopic ventral hernia repair surgery.

DETAILED DESCRIPTION:
Ventral hernia repair is a very common surgical operation. Both laparoscopic and robot-assisted operations are considered acceptable. However, there is no clear indication for a particular approach. No prospective trial has been conducted so far to establish superiority of one approach over the other. The Investigator believes each approach has unique characteristics and may offer advantages over the other in the right population group. The Investigator will randomly assign patients in two arms according to the surgical approach, whether laparoscopic or robot-assisted. The Investigator will collect preoperative characteristics, intraoperative variables, and postoperative outcomes. The Investigator will compare all variables to establish differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* surgeon determined need for ventral hernia repair

Exclusion Criteria:

* <18 & >99 years of age
* Pregnant
* Medical indication for open repair

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Operative time | perioperative time
  time from start to finish of procedure, procedure start and stop times as recorded by anesthesia

SECONDARY OUTCOMES:
Post operative pain score | until year five post-operative
  Abdominal pain at rest and on moving (recumbent to the upright position), will be assessed using 0-10 Numeric Pain Rating Scale preoperatively (baseline), and at 24 hours, 30 days, and one year postoperatively

OTHER OUTCOMES:
Complications | From immediately post-operative until year five following surgical ventral hernia repair.
  Post-operative 30 day complication rates will be recorded prospectively. All complications (including multiple occurrences per patient) will be recorded and graded per the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Latzko, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States